CLINICAL TRIAL: NCT04601909
Title: A Phase 1b, Prospective, Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Multicenter, Safety Study of FX-322 Administered by Intratympanic Injection in Adults With Age-Related Sensorineural Hearing Loss
Brief Title: FX-322 in Adults With Age-Related Sensorineural Hearing Loss
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Frequency Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX-322-112
Record Dates: First submitted 2020-10-12; First posted 2020-10-26 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Presbycusis; Hearing Loss, Sensorineural; Noise Induced Hearing Loss; Sudden Hearing Loss
Keywords: Intratympanic administration; Restoration of hearing loss
MeSH Terms: conditions — Presbycusis; Hearing Loss, Sensorineural; Hearing Loss, Noise-Induced; Hearing Loss, Sudden

STUDY DESIGN:
Intervention Model Description: Approximately 30 subjects are planned to be enrolled in this study. The subjects will be randomized to receive FX-322 or placebo randomized 4:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FX-322 (Active Comparator): FX-322, 1 dose (N=24)
  Interventions: Drug: FX-322
- Placebo (Placebo Comparator): Placebo, 1 dose (n=6)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: FX-322 — active comparator
  Arms: FX-322
Other: placebo — placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1b, prospective, randomized, double-blind, placebo-controlled, single-dose, multicenter, safety study of FX-322, administered by intratympanic injection, in adults with age-related sensorineural hearing loss.

DETAILED DESCRIPTION:
This is a Phase 1b placebo-controlled, double-blind, randomized, single-dose safety study of intratympanic FX-322 dosed in subjects with age-related sensorineural hearing loss.

Approximately 30 subjects are planned to be enrolled in this study. The subjects will be randomized to receive one dose FX-322 (24) or placebo (6) and will return for safety, otologic, and audiologic assessments at Days 30 and 90 after the study injection.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has read and voluntarily signed the Informed Consent Form (ICF) after all questions have been answered and prior to any study-mandated procedure.
2. Adult aged 66-85 years inclusive.
3. Documented medical history consistent with age-related sensorineural hearing loss (documented audiogram at least 6 months prior to screening required).
4. A pure tone average of 26-70 dB at 500Hz, 1000Hz, 2000Hz, and 4000Hz at Screening in the ear to be injected.
5. Ability to communicate well with the Investigator and is willing to comply with and complete all the study procedures.

Exclusion Criteria:

1. Subject has previously participated in a FX-322 clinical trial.
2. Any subject with a flat audiogram between 500Hz and 8000Hz at Screening in the study ear. The difference in the range of threshold values across frequencies is ≤15 dB for the definition of a flat audiogram.
3. Clinically significant abnormalities on safety laboratory tests.
4. Perforation of tympanic membrane or other tympanic membrane disorders that would interfere with the delivery and safety assessment of an intratympanic medication or reasonably be suspected to affect tympanic membrane healing after injection in study ear. This includes a current tympanostomy tube.
5. Any conductive hearing loss of greater than 15 dB at a single frequency or greater than 10 dB at two or more contiguous octave frequencies in the study ear at the Screening visit or on the prior audiogram (if the Investigator feels there is not a true conductive hearing loss, the Medical Monitor should be consulted).
6. Active chronic middle ear disease or a history of major middle ear surgery, as an adult, in the ear to be injected.
7. Subject has had an intratympanic injection in either ear within 3 months of the screening visit.
8. History of clinically significant vestibular symptoms at the discretion of the investigator. For example, BPPV may be considered acceptable whereas Meniere's would not.
9. History of clinically significant systemic autoimmune disease (e.g. rheumatoid arthritis, Sjogren's syndrome, multiple sclerosis, psoriasis).
10. Exposure to another investigational drug within 28 days prior to injection of study drug.
11. Evidence of any active or chronic disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would pose an unacceptable risk to the subject in the opinion of the investigator following a detailed medical history, physical examination, and vital signs (systolic and diastolic blood pressure, pulse rate, body temperature).
12. Females of childbearing potential (those who are not surgically sterilized or post-menopausal) may not participate in the study if any of the following conditions exist:

    * Pregnant or intend to become pregnant
    * Nursing (lactating)
    * Does not agree to use adequate birth control methods for the duration of the study (adequate birth control methods are: hormonal- oral, implantable, transdermal or injectable contraceptives; mechanical- spermicide in conjunction with a barrier such as a condom or diaphragm, IUD, or surgical sterilization of a partner.

    NOTE: all female subjects of childbearing potential must consent to a urine pregnancy test as described in the Schedule of Assessments
13. Any known factor, condition, or disease that, in the view of the Investigator, might interfere with treatment compliance, study conduct or interpretation of the results (e.g. previous high-dose aminoglycoside treatment).

Ages: 66 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Systemic Safety: Number of patients with treatment-related adverse events | 3 months
  Number of patients with treatment-related adverse events assessed by CTCAE v5.0
Local Safety: Number of patients with abnormal changes from baseline in otoscopic examinations | 3 months
  Microscopic otoscopy will be included to specifically record any abnormalities of the external ear canal, tympanic membrane and middle ear.
Local Safety: The number of patients with abnormal changes from baseline in tympanometry | 3 months
  Tympanometry tests the integrity of the tympanic membrane by varying air pressure in the ear canal. Middle ear compliance (mL), peak pressure (daPa), and ear canal volume (mL) will be recorded.
Columbia-Suicide Severity Rating Scale (C-SSRS) | 3 months
  Risk assessment through a series of simple, plain-language questions

SECONDARY OUTCOMES:
Audiologic Response Endpoints: Speech Intelligibility - Word Recognition in Quiet (WR) | 3 months
  Assessment of speech intelligibility using the Word Recognition in Quiet test measured with Consonant-Nucleus-Consonant (CNC) word lists.
Audiologic Response Endpoints: Speech Intelligibility - Words-In-Noise (WIN) | 3 months
  Speech intelligibility using the Words-in-Noise test measured with Consonant-Nucleus-Consonant (CNC) word lists
Standard Pure Tone Audiometry | 3 months
  Standard pure tone audiometry will be measured to determine a subject's threshold for hearing at standard frequencies (Hz)
Extended High Frequency Pure Tone Audiometry | 3 months
  Pure tone audiometry will be measured to determine a subject's threshold for hearing at extended high range frequencies (Hz)
Tinnitus Assessment | 3 months
  Measured by the Tinnitus Functional Index (TFI), with a scale ranging from 0 to 100 that defines severity categories based on 25 self-reported answers.

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Director — Frequency Therapeutics
Locations (5):
- United States (5):
  - Clinical Trial Site, Sarasota, Florida
  - Clinical Trial Site, Omaha, Nebraska
  - Clinical Trial Site, Amherst, New York
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No